CLINICAL TRIAL: NCT03659318
Title: Is Clinical Outcome of Robotic-Assisted TKA Better Than Conventional Manual TKA?Prospective, Randomized Study
Brief Title: Robotic-Assisted Versus Conventional Total Knee Arthroplasty(TKA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, Young Hoo Kim, Professor, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RoboTKA
Record Dates: First submitted 2018-08-19; First posted 2018-09-06 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Arthritis; Knee Arthropathy; Robotics
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot (Experimental): TKA is done with robotic-assisted manner. Final implantation of implants is done by surgeons, same as the conventional way. Robotic-assisted TKA for this arm.
  Interventions: Procedure: Robotic-assisted TKA
- Conventional (Active Comparator): TKA is done with conventional instruments. Conventional TKA for this arm.
  Interventions: Procedure: Conventional TKA

INTERVENTIONS:
Procedure: Robotic-assisted TKA — Total knee arthroplasty is carried out with help of robotic surgery system, using a Robodoc system. CT-based preoperative planning using ORTHODOC (Integrated Surgical Technology Corp) performed in the first step before the day of surgery, and the robotic-assisted surgery using the ROBODOC surgical assistance in the second step. The bone markers are registered to the computer, and the computer arm does all the cutting and preparation of bones. This is in contrast to conventional jigs and cutting blocks. Actual implantation of the implants is done by a surgeon. A Duracon posterior cruciate-substituting total knee prosthesis (Stryker Orthopedics, Mahawh, NJ, USA) are used in all knees.
  Arms: Robot
Procedure: Conventional TKA — Total knee arthroplasty is carried out with classical, conventional, manual method. A surgeon measures the angle, length of the cuts with bone landmarks and specialized surgical instruments. After all the cuts actual implantation is done. A Duracon posterior cruciate-substituting total knee prosthesis (Stryker Orthopedics, Mahawh, NJ, USA) are used in all knees.
  Arms: Conventional

SUMMARY:
Robotic-assisted total knee arthroplasty (TKA) was introduced to attempt to enhance the precision of bone preparation, component alignment and ultimately improve clinical results and survivorship of TKA. Although several published data suggest that bone preparation, and knee component alignment were improved by using robotic assistance, there is no high-quality evidence from randomized trials at long-term of which investigators are aware evaluating whether the improved bone preparation and knee component alignment improved clinical function or longevity of the TKA.

DETAILED DESCRIPTION:
Robotic-assisted TKA was introduced in an attempt to enhance component alignment and to improve long-term clinical results and implant durability, particularly in younger patients. Several comparative studies of conventional and robotic-assisted TKAs demonstrated that improved alignment of the components was obtained after the robotic-assisted TKAs than conventional TKAs.

To date, however, no comprehensive synthesis of long-term randomized data has been conducted specifically for robotic-assisted TKA, particularly in younger patients. It is crucial to determine whether improved alignment of the TKA components obtained by using robotic-assistance, would improve better long-term and functional results and survivorship of TKAs.

The aims of the current study were to examine the two groups of patients after long-term follow-up to determine whether the clinical results, radiographic and CT scan results, and the survivorship of TKA would be better after robotic-assisted TKA than after conventional TKA.

ELIGIBILITY:
Inclusion Criteria:

* end stage knee arthritis

Exclusion Criteria:

* mild knee deformity
* inflammatory arthritis
* foot and ankle disorder
* dementia
* hip disease
* history of a stroke
* older than 65 years of age

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 674 (Actual)
Dates: Start 2002-01 (Actual); Primary Completion 2008-02 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Knee society Knee score | 20 years after the surgery
  a proven score for the measurement of knee function, the score ranges from 0 to 100, 100 being the best possible score, indicating normal knee function

SECONDARY OUTCOMES:
WOMAC score | 20 years after the surgery
  A tool to evaluate patient function associated with knee. The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). The total score is summed from individual sections, and 0 is the best possible score.

REFERENCES:
- [Background] Arima J, Whiteside LA, McCarthy DS, White SE. Femoral rotational alignment, based on the anteroposterior axis, in total knee arthroplasty in a valgus knee. A technical note. J Bone Joint Surg Am. 1995 Sep;77(9):1331-4. doi: 10.2106/00004623-199509000-00006. PMID 7673281
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Bellemans J, Vandenneucker H, Vanlauwe J. Robot-assisted total knee arthroplasty. Clin Orthop Relat Res. 2007 Nov;464:111-6. doi: 10.1097/BLO.0b013e318126c0c0. PMID 17563698
- [Background] Crowder AR, Duffy GP, Trousdale RT. Long-term results of total knee arthroplasty in young patients with rheumatoid arthritis. J Arthroplasty. 2005 Oct;20(7 Suppl 3):12-6. doi: 10.1016/j.arth.2005.05.020. PMID 16213997
- [Background] Decking J, Theis C, Achenbach T, Roth E, Nafe B, Eckardt A. Robotic total knee arthroplasty: the accuracy of CT-based component placement. Acta Orthop Scand. 2004 Oct;75(5):573-9. doi: 10.1080/00016470410001448. PMID 15513489
- [Background] Jacofsky DJ, Allen M. Robotics in Arthroplasty: A Comprehensive Review. J Arthroplasty. 2016 Oct;31(10):2353-63. doi: 10.1016/j.arth.2016.05.026. Epub 2016 May 18. PMID 27325369